CLINICAL TRIAL: NCT02132975
Title: Pilot Study of a Motorised Probe Holder Assisting Prostate Biopsies
Brief Title: Motorised Probe Holder Assisting Prostate Biopsies
Acronym: PROSBOT-Apollo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdministrateurCIC (Other)
Collaborators: Pitié-Salpêtrière Hospital (Other); Institute for Intelligent Systems and Robotics (Unknown); Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor-Investigator, AdministrateurCIC, Coordinating investigator, University Hospital, Grenoble
Organization: University Hospital, Grenoble (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DCIC 14 05
Record Dates: First submitted 2014-04-25; First posted 2014-05-07 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With motorised probe handler (Experimental): The surgeon use the motorised probe handler to do the biopsy
  Interventions: Device: Biopsies using Apollo and UroStation®; Procedure: Biopsies using UroStation® (image fusion)
- Without motorised probe handler (Experimental): The surgeon do the biopsy as he usually do.
  Interventions: Procedure: Biopsies using UroStation® (image fusion)

INTERVENTIONS:
Device: Biopsies using Apollo and UroStation® — Apollo : Motorised probe handler for prostate biopsies
  Arms: With motorised probe handler
Procedure: Biopsies using UroStation® (image fusion)

SUMMARY:
Study, for the first time in clinical conditions, the potential contribution, in terms of accuracy, of the motorised probe holder during prostate biopsies.

ELIGIBILITY:
Inclusion Criteria:

* of-age patient
* patient for whom a prostate biopsies session is planned
* patient affiliated to the social security or equivalent
* patient having a target identified on MRI
* Written informed consent

Exclusion Criteria:

* contraindication
* patient wearing a mechatronic device
* patient concerned by the L1121-6 à 8 of the health public code

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Distance between virtual and effective biopsy, in the two arms | 8 months

SECONDARY OUTCOMES:
Success rate in locking/releasing the probe combined with success rate in performing a full exploration of the prostate | 8 months
Probe holder positions error between virtual and effective biopsy | 8 months
User satisfaction | 2 hours
  * biopsies session duration
  * device manageability
  * device unwiediness
  * contribution of the lock of the probe
  * set up, cleaning
  * global satisfaction
Safety Evaluation | 2 hours
  * number of time the device couldn't be started
  * number of times the emergency button was pushed
  * number of time the biopsy couldn't entirely be done using the device
  * number of time the device protections had to be repositioned

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Mozer, MD, PhD, Principal Investigator — AP-HP Pitié Sapêtrière
Locations (1):
- Urology, AP-HP Pitié Salpêtrière, Paris, Île-de-France Region, France

REFERENCES:
- See also: Related Info — http://www.cic-it-grenoble.fr/